CLINICAL TRIAL: NCT00779987
Title: Autologous Serum Efficacy Study in Patients With Severe Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Cristhian A Urzua, University of Chile
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP261
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2008-10

CONDITIONS: Dry Eye
Keywords: Dry eye; Autologous serum; Ocular Surface Disease Index
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous serum -Systane (Other): Crossover arm starting with autologous serum for 2 weeks. After a 1 week wash out with 0.9% sodium chloride, they continue with 2 weeks using artificial tears (Systane)
  Interventions: Drug: Autologous serum - Systane
- Systane- Autologous serum (Other): Crossover arm starting with artificial tears (Systane) for 2 weeks. After a 1 week wash out with 0.9% sodium chloride, they continue with 2 weeks using autologous serum.
  Interventions: Drug: Systane - Autologous serum

INTERVENTIONS:
Drug: Autologous serum - Systane — 20% autologous serum solution used four times a day for two weeks. Then 0.9% sodium chloride four times a day for one week. Finally, Systane (r) four times a day for two weeks.
  Arms: Autologous serum -Systane
Drug: Systane - Autologous serum — Systane (r) four times a day for two weeks. Then 0.9% sodium chloride used four times a day for one weeks. Finally, 20% autologous serum solution four times a day for two week.
  Arms: Systane- Autologous serum

SUMMARY:
The purpose of this study is to compare the reduction in symptomatology of patients with severe dry eye treated with autologous serum and conventional artificial tears.

DETAILED DESCRIPTION:
Severe dry eye remains an important and frequent eye disease, that reflects in a severe impairment of the patient´s life quality. Up to date there is no ideal therapy for this condition. Few studies have reported some kind of improvement in different parameters related to dry eye with the use of autologous serum, but no one has considered the patient´s symptoms with a systematic and validated evaluation method.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Severe Dry Eye, as defined by a OSDI score > or = 40

Plus:

* Tear Break Up Time (TBUT) < 5 seconds
* Cornea-conjunctival epithelial defects measured by Fluorescein staining and evaluation using the Oxford score.

Exclusion Criteria:

* No dry eye associated ocular disease
* Unable to comply protocol
* Severe anemia
* Previous use of autologous serum
* Concomitant use of other topical ocular drug
* Hypersensibility to any proposed interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To compare the score reduction in the Ocular Surface Disease Index (OSDI) between patients treated with autologous serum and conventional artificial tears. | 5 weeks

SECONDARY OUTCOMES:
To compare variations in objective eye measurements, such as Tear Break Up Time and corneal-conjunctival staining according to the Oxford Score, in patients treated with autologous serum and conventional artificial tears. | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cristhian A Urzua, MD, Principal Investigator — University of Chile
Locations (1):
- University Of Chile Clinical Hospital, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Derived] Urzua CA, Vasquez DH, Huidobro A, Hernandez H, Alfaro J. Randomized double-blind clinical trial of autologous serum versus artificial tears in dry eye syndrome. Curr Eye Res. 2012 Aug;37(8):684-8. doi: 10.3109/02713683.2012.674609. Epub 2012 Jun 6. PMID 22670856